CLINICAL TRIAL: NCT02840123
Title: Phase Ib Clinical Trial on the Safety of Immunotherapy With Autologous Dendritic Cells Primed With Lysate Allogeneic Tumor Lines in Patients With Diffuse Intrinsic Pontine Glioma (DIPG)
Brief Title: Safety Study of DIPG Treatment With Autologous Dendritic Cells Pulsed With Lysated Allegenic Tumor Lines
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSJD-DIPG-DC
Record Dates: First submitted 2016-05-31; First posted 2016-07-21 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

ARMS (1):
- Autologous dendritic cells (Experimental)
  Interventions: Biological: Autologous dendritic cells

INTERVENTIONS:
Biological: Autologous dendritic cells

SUMMARY:
The purpose of this study is to asses safety of diffuse intrinsic pontine glioma (DIPG) treatment with autologous dendritic cells pulsed with lysated allegenic tumor lines

Evaluate the nonspecific immune response generated in peripheral blood and Cerebral Spinal Fluid (CSF) by proposed treatment Evaluate the specific antitumor immunity response generated in peripheral blood and CSF Assess overall survival and progression free survival Correlate the neuroradiological changes with the clinical course and immune response generated in peripheral blood and CSF Quality of life evaluation

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed DIPG Patients without progressive disease
* Aged between 3 and 18 yo Lansky scale >50 (Karnofsky for patients aged more than 16 yr)
* Life expectancy > 8 weeks
* Preserved bone marrow function Normal hepatic and renal function

Exclusion Criteria:

* Impossibility to perform aphaeresis
* Patient participation of other experimental study within the last 3 months
* Patient under antitumor treatment in the last 4 weeks
* Co-morbidity that does not allow the study treatment
* Patients requiring > 2mg/day of dexamethasone treatment Corticoid-dependent patients
* Patients under uncontrolled infection
* Positive serologies of HIV, hepatitis C virus (HCV) or hepatitis B virus (HBV)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events per patient (after treatment administration | 2 years

SECONDARY OUTCOMES:
Overall survival Progression free survival | 1 year
Time to first Serious Adverse Event (SAE)(after treatment) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain